CLINICAL TRIAL: NCT00534209
Title: Phase I/II Clinical Trial of Immunotherapy With an Allogeneic B7.1/HLA-A1 Transfected Tumor Cell Vaccine in Patients With Stages IIIB/IV Non-Small Cell Lung Cancer That Have Completed First Line Chemotherapy
Brief Title: Vaccine Therapy in Patients With Stages IIIB/IV Non-Small Cell Lung Cancer Who Have Finished First-Line Chemotherapy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Per request of Principal Investigator this study was closed.
Sponsor: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20057158; SCCC-2005042 (Other: UM/Sylvester Comprehensive Cancer Center); WIRB-20051678 (Other: Western IRB (WIRB))
Record Dates: First submitted 2007-09-20; First posted 2007-09-24 (Estimated); Results first posted 2013-02-20 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-09

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — B7-1 Antigen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I: Allogeneic B7.1/HLA-A1 (Experimental): Patients will receive Allogeneic B7.1/HLA-A1 vaccine once every other week for 2 courses over 12 weeks, for a maximum of 6 vaccines.
  Given intradermally.
  Interventions: Biological: Allogeneic B7.1/HLA-A1
- Arm II: Placebo (Placebo Comparator): Patients receive a placebo vaccine intradermally once every other week for 2 courses over 12 weeks, for a maximum of 6 vaccines.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Allogeneic B7.1/HLA-A1 — Dose: At least 4x10^7 irradiated HLA/B7.1 transfected AD100 cells Given intradermally
  Other Names: - B7.1; - B7; - Ad100-B45-Neo-B7.1-HLA A1 or HLA2
  Arms: Arm I: Allogeneic B7.1/HLA-A1
Other: Placebo — Given intradermally
  Arms: Arm II: Placebo

SUMMARY:
RATIONALE: Vaccines made from gene-modified tumor cells may help the body build an immune response to kill tumor cells.

PURPOSE: This randomized phase I/II trial is studying the side effects of vaccine therapy and to see how well it works in treating patients with stage IIIB or stage IV non-small cell lung cancer who have finished first-line chemotherapy.

DETAILED DESCRIPTION:
OUTLINE: This is a multicenter study.

* Phase I (single site [University of Miami Sylvester Comprehensive Cancer Center]): Patients receive allogeneic B7.1 and human leukocyte antigen-A1 (HLA-A1) transfected tumor cell vaccine intradermally (ID) in weeks 1, 3, and 5. Treatment repeats every 6 weeks for 2 courses. If no more than 1 of 6 patients experience a probable or definitively treatment related adverse effect (i.e., grade 2 autoimmune or grade 3-4 of any type), patients proceed to the phase II portion of the study. If 2 or more (out of 6) patients experience treatment related adverse effects the study stops.
* Phase II (randomized): Patients are stratified according to study site (University of Miami Sylvester Comprehensive Cancer Center or Memorial Regional Hospital), type of prior first-line treatment (platinum and taxane vs platinum and gemcitabine), and presence of brain metastasis (yes vs no). Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive allogeneic B7.1 and HLA-A1 transfected tumor cell vaccine ID in weeks 1, 3, and 5. Treatment repeats every 6 weeks for 2 courses.
  * Arm II: Patients receive a placebo vaccine as in arm I. Patients undergo blood sample collection periodically for correlative studies. Samples are analyzed for cluster of differentiation 8 (CD8), cluster of differentiation 4 (CD4), and natural killer cell (NK) response and peripheral blood lymphocytes (PBL) and T helper cell 1 (TH1)/T helper cell 2 (TH2) bias, including levels of interleukin (IL) IL-1β, IL-2, IL-4, IL-5, IL-6, IL-13, Interferon-gamma (IFN-γ), tumor necrosis factor-alpha (TNF-α) via ELISA.

After completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 4 years, and then once a year thereafter.

PROJECTED ACCRUAL: A total of 66 patients (6 patients for phase I and 60 patients for phase II) will be accrued for this study.

ELIGIBILITY:
INCLUSION CRITERIA

* Patients with stage IIIB (non-candidates for radiation) or stage IV pathologically confirmed non-small cell carcinoma of the lung that completed 4-6 cycles of platinum based first line chemotherapy and achieved complete response (CR), partial response (PR) or stable disease.
* Last administration of chemotherapy occurred no later than 4 weeks prior to the enrollment date.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Renal Requirements: The calculated creatinine clearance must be at least 50 ml/min.
* Pulmonary Function Requirements:

  * All patients will undergo evaluation of pulmonary function prior to enrollment.
  * Patients should have a Forced expiratory volume in 1 second (FEV1) more than 30% of the predicted value and/or Diffusing capacity (DLCO) more than 30% of the predicted value with a partial pressure of carbon dioxide (PCO2) < 45mm.
  * Any patient enrolled in the protocol whose respiratory symptoms have experienced marked deterioration not related to a known cause (e.g. pneumonia, congestive heart failure (CHF) or pulmonary embolism (PE)) will have request pulmonary function test (PFT) evaluation and if the above parameters are seen will be excluded from the protocol.
* Age ≥ 18 years.
* Signed informed consent.
* Patients should have absolute neutrophil count (ANC) ≥ 1000/mm3; platelets (PLT) ≥ 80,000/mm3.

EXCLUSION CRITERIA:

* Small cell carcinoma of the lung.
* Existing autoimmune disorders such as rheumatoid arthritis, systemic lupus erythematosus, Sjogren's disease etc; colitis, inflammatory bowel disease or pancreatitis within 10 years of study.
* Other active malignancies present within the past three years, except for basal and/or squamous cell carcinoma(s) or in situ cervical cancer.
* Concomitant steroid or other immunosuppressive therapy.
* Active infection, or less than 7 days since therapy for acute infections.
* Pericardial effusion.
* Currently receiving chemotherapy for another condition (such as arthritis).
* Time elapsed greater than 4 weeks since last administration of first line chemotherapy for NSCLC.
* Active or symptomatic cardiac disease such as congestive heart failure, angina pectoris or recent myocardial infarction.
* Pregnant or lactating women (negative test for pregnancy required of women of childbearing potential).
* Refusal in fertile men or women to use effective birth control measures during and for six months after the completion of treatment on study.
* Known HIV infection
* Untreated or uncontrolled brain metastasis.
* Liver Enzymes greater than 3 times the institutional upper limit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luis E. Raez, MD, FACP, Study Chair — University of Miami Sylvester Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Memorial Regional Hospital, Hollywood, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida

REFERENCES:
- [Background] Raez LE, Cassileth PA, Schlesselman JJ, Padmanabhan S, Fisher EZ, Baldie PA, Sridhar K, Podack ER. Induction of CD8 T-cell-Ifn-gamma response and positive clinical outcome after immunization with gene-modified allogeneic tumor cells in advanced non-small-cell lung carcinoma. Cancer Gene Ther. 2003 Nov;10(11):850-8. doi: 10.1038/sj.cgt.7700641. PMID 14605671
- [Background] Frankowski DJ, Raez J, Manners I, Winnik MA, Khan SA, Spontak RJ. Formation of dispersed nanostructures from poly(ferrocenyldimethylsilane-b-dimethylsiloxane) nanotubes upon exposure to supercritical carbon dioxide. Langmuir. 2004 Oct 12;20(21):9304-14. doi: 10.1021/la049646l. PMID 15461522

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I: Patients will receive B7 vaccine once every other week for 2 courses over 12 weeks, for a maximum of 6 vaccines.
  Given intradermally.
Period: Overall Study
Arm/Group | Arm I
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm I
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Preliminary Safety Profile (Phase 1)
Description: This will include the number of patients experiencing toxicity over the course of treatment, characterized by type of toxicity and grade, and by the time of toxicity onset in relation to day of vaccination.
Time Frame: Up to 13 weeks
Measure: Number; unit: participants
Arm/Group | Arm I
Number analyzed (Participants) | 1
participants | 1

2. Primary Outcome: Progression-free Survival (Phase 2)
Time Frame: Date of randomization to the earliest date of documented progression.
Population: This was an outcome measure for the Phase 2 portion of the study, which was never opened to accrual. No participants were enrolled in Phase 2 therefore no data were available.
Groups:
- Arm I: Allogeneic B7.1/HLA-A1: Patients will receive Allogeneic B7.1/HLA-A1 vaccine once every other week for 2 courses over 12 weeks, for a maximum of 6 vaccines.
  Given intradermally.
  Allogeneic B7.1/HLA-A1: Dose: At least 4x10^7 irradiated HLA/B7.1 transfected AD100 cells Given intradermally
Arm/Group | Arm I: Allogeneic B7.1/HLA-A1 | Arm II: Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Immune Response (CD8) in B7-vaccinated Participants as Compared to Controls. (Phase 2)
Description: Rate of immune response (CD8) in B-7 vaccinated participants reported for measurements taken immediately prior to vaccination (week 0) and throughout the two courses.
Time Frame: About 13 weeks
Population: as for outcome 2
Arm/Group | Arm I: Allogeneic B7.1/HLA-A1 | Arm II: Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Relationship of CD8 Response in B7-vaccinated Patients to Their Progression-free Survival.(Phase 2)
Description: Relationship of CD8 response in B7-vaccinated patients to their progression-free survival. Summarized by the median and range of follow up time for patients grouped according to disease status (progression/no progression) and vital status (died/alive at last contact).
Time Frame: From Week 1 of Study Therapy until Death or Withdrawal of Consent
Population: as for outcome 2
Arm/Group | Arm I: Allogeneic B7.1/HLA-A1 | Arm II: Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Safety Profile (Phase 2)
Description: The rate of patients experiencing toxicity over the course of treatment will be characterized by type of toxicity and grade, and by the time of toxicity onset in relation to day of vaccination.
Time Frame: About 13 weeks
Population: as for outcome 2
Arm/Group | Arm I: Allogeneic B7.1/HLA-A1 | Arm II: Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Response to Second-line Chemotherapy After Disease Progression (Phase 2)
Description: The percentage of patients experiencing a clinical response (complete response (CR), partial response (PR), stable disease (SD)) on second-line chemotherapy will be characterized for B7-vaccinated patients and controls.
Time Frame: From Week 1 of Study Therapy until Death or Withdrawal of Consent
Population: as for outcome 2
Arm/Group | Arm I: Allogeneic B7.1/HLA-A1 | Arm II: Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Overall Survival (Phase 2)
Description: The length of time from either the date of diagnosis or the start of treatment for a disease, such as cancer, that study participants are still alive.
Time Frame: Date of randomization to the recorded date of death
Population: as for outcome 2
Arm/Group | Arm I: Allogeneic B7.1/HLA-A1 | Arm II: Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Correlative Immunological Studies in Study Participants (Phase 2)
Description: The time course of patients' adaptive immune response to B7 vaccination as compared to control vaccine will be characterized by their CD8, CD4, and NK response (measured by ELI-spots for interferon-gamma (IFN-γ), interleukin 4 (IL-4), and granzyme B secretion) measured prior to vaccination (i.e. at baseline) and over two courses of vaccination (measurements at week 7 and 13).
Time Frame: Baseline, Week 7 and Week 13
Population: as for outcome 2
Arm/Group | Arm I: Allogeneic B7.1/HLA-A1 | Arm II: Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm I
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=1)
Grade 3 Edema limbs (Musculoskeletal and connective tissue disorders) | 1 (1)
Grade 3 Vascular access complication (Blood and lymphatic system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study closed early due to low enrollment. A minimum of 2 patients were required for Phase 1, however, this requirement was not met.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes